CLINICAL TRIAL: NCT04374266
Title: Clinical and Postoperative Radiologic Assessment and Long Term Results of Tegmen Defects During Mastoidectomy
Brief Title: Tegmen Defect Management During Mastoidectomy
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, ahmet mutlu, Dr, Istanbul Medeniyet University
Other Study IDs: Tegmen defect
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Chronic Otitis Media
MeSH Terms: interventions — Physical Examination; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: physical examination, and computerized tomography — physical examination, and computerized tomography was performed during routine follow-up

SUMMARY:
In this study, we aimed to discuss our clinical experience on the management of the tegmen defects which were revealed during the mastoidectomy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* underwent mastoidectomy as alone or as a part of the surgery, and noticed tegmen mastoideum or tympani defect in related department.

Exclusion Criteria:

* patients who did not come to follow up

Ages: 12 Years to 74 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: underwent mastoidectomy as alone or as a part of the surgery, and noticed tegmen mastoideum or tympani defect in related department.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
defect size | a year
  decreased size of the defects were examined

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided